CLINICAL TRIAL: NCT04262037
Title: A Comparative Study of Three Modes of Ventilation During Cardiopulmonary Bypass in Pediatric Patients With Pulmonary Hypertension Undergoing Congenital Heart Disease Surgeries
Brief Title: A Comparative Study of Three Modes of Ventilation During CPB in Pediatrics With Pulmonary Hypertension Undergoing Congenital Heart Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Madkour, Lecturer of Anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N-12/2019 MD
Record Dates: First submitted 2019-08-13; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Congenital Heart Disease; Pulmonary Hypertension
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HPPV (Experimental): will receive high frequency positive pressure ventilation during cardiopulmonary bypass at tidal volume 2 ml/kg and respiratory rate 80. Lung ultrasound will be done at the beginning and end of surgery
  Interventions: Diagnostic Test: lung ultrasound
- CPPV (Experimental): will receive continuous positive airway pressure of 10 cmH2o during the bypass. Lung ultrasound will be done at the beginning and end of surgery
  Interventions: Diagnostic Test: lung ultrasound
- Control (No Intervention): will be disconnected from the ventilation (passive deflation). Lung ultrasound will be done at the beginning and end of surgery.Lung ultrasound will be done at the beginning and end of surgery

INTERVENTIONS:
Diagnostic Test: lung ultrasound — Lung ultrasound will be performed after induction of anesthesia and at the end of the operation with a 5-MHz curved array probe (MindrayDC-N6; Mindray; Shenzhen, China
  Arms: CPPV; HPPV

SUMMARY:
Aim of Work:

The aim of this randomized, double-blinded, study is to compare between three modes of ventilation during cardiopulmonary bypass in pediatric patients with pulmonary hypertension undergoing corrective cardiac surgeries.

Hypothesis:

The hypothesis of the present study is that high frequency low volume positive pressure ventilation is better than continous positive airway pressure (CPAP)and passive deflation on direct PAP (pulmonary artery pressure ) reading and immediate oxygenation after cardiopulmonary bypass CPB in pediatric patients undergoing cardiac surgeries for congenital heart defects.

DETAILED DESCRIPTION:
The patients will be randomized in a double blinded fashion to get enrolled into 3 equal groups: Group HFPPV patients (n = 8) will receive high frequency positive pressure ventilation during cardiopulmonary bypass at tidal volume 2 ml/kg and respiratory rate 80, whereas Group CPPV patients (n = 8 ) will receive continuous positive airway pressure of 10 cmH2O during the bypass, while Control group patients (n = 8 ) will be disconnected from the ventilation (passive deflation) .The study will be conducted in the pediatric cardio-thoracic operation rooms in AbulReesh Hospital in Cairo University.

Advanced Monitoring where Naso-pharyngeal temperature probe will be placed, a Central venous catheter to monitor central venous pressure and an arterial cannula to monitor invasive blood pressure after that, standard cardiopulmonary bypass technique will be used in all patients. Before aortic cannulation, patients will receive IV heparin 400 U.kg-1 aiming to produce activated clotting time ACT value > 400 sec. A membrane oxygenator (minimax plus; Medtronics Inc.) will be used during cardiopulmonary bypass. Priming solution in the form of iso-tonic saline solution supplemented with heparin added to fresh whole blood in appropriate amounts to achieve a haematocrit 20-25% during CPB will be used. Furosemide in a dose of 1 mg/kg/min will be given to all patients. Venting of left heart will be performed with a left atrial vent inserted through a small incision at the inter-atrial septum. Anesthesia during CPB will be given by Sevoflurane administrated via a vaporizer inserted into the oxygenator gas supply with a constant gas flow 3 liter/min. A non-pulsatile roller pump (model10.10.00; Stocket instruments; Munich, Germany) will be used and the pump flow will be adjusted at 2.4 to 2.6 L/min /m2 during the normothermic period targeting mean arterial blood pressure between 40 and 60 mmHg. Moreover, all patients will receive milrinone loading dose of 50mcg/kg/min the maintanence 0.5-1 mcg/kg/min and or adrenaline 0.02-0.1 mcg/kg/min will be utilized to facilitate weaning from CPB.

After sternotomy and direct exposure of the pulmonary artery, the pulmonary artery systolic pressure (PASP) will be monitored by a direct arterial catheter 22 gauge inserted by the surgeon into the pulmonary artery, was calculated and recorded immediately after sternotomy, after aortic clamp removal, and 10 minutes after initiation of protamine infusion).

After application of aortic cross clamp and administration of cold blood cardioplegia solution (Saint Thomas cardioplegic solution) 40 ml/Kg to be followed by doses of 10ml/Kg every 30 minutes.), Group A patients will receive high frequency low volume positive pressure ventilation (HFPPV) during cardiopulmonary bypass at tidal volume Vt 2 ml/kg and respiratory rate RR 80, whereas Group B patients (n =8 ) will receive continous positive airway pressure CPAP of 10 cmH2O, and group C patients will be disconnected from the ventilator (passive deflation) .

Finally, Lung Ultrasound Score will be obtained after induction of anesthesia and at the end of surgery after chest closure, The duration of mechanical ventilation, length of stay in the intensive care unit and immediate post bypass oxygenation as well as the requirement for inotropic and vaso-tropic support during the first 24 hours study period will be recorded for all patients

Lung ultrasound protocol:

Lung ultrasound will be performed after induction of anesthesia and at the end of the operation with a 5-MHz curved array probe (MindrayDC-N6; Mindray; Shenzhen, China). Patients will be investigated in supine position by a well-trained physician recording five seconds videos that will be assessed by two different observers who will be blinded from the patient data. Lung ultrasound will be assessed for the presence of B lines.

ELIGIBILITY:
Inclusion Criteria:

* Age: 4 months to 6 years.
* ASA I, II, III.
* Patients undergoing atrial septal defect or ventricular septal defect or common atrio-ventricular canal corrective cardiac surgeries on cardiopulmonary bypass
* Patients suffering moderate to severe pulmonary hypertension.

Exclusion Criteria:

* Any congenital anomalies of the lung as cystic fibrosis, congenial diaphragmatic hernia.
* ASA IV.
* Mild pulmonary hypertension or normal PAP.
* Patients who will require high doses of inotropes (adrenaline > 0.1 mcg/kg/min or milrinone > 1 mcg/kg/min) will be excluded from the study.

Ages: 4 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
• Direct pulmonary artery systolic pressure (PASP) measured in mmHg | immediately after sternotomy,
  the pulmonary artery systolic pressure (PASP) will be monitored by a direct arterial catheter 22 gauge inserted by the surgeon into the pulmonary artery, immediately after sternotomy, after aortic clamp removal, and 10 minutes after initiation of protamine infusion
Change in direct pulmonary artery systolic pressure (PASP) measured in mmHg | after aortic clamp removal 10 minutes after initiation of protamin
  the pulmonary artery systolic pressure (PASP) will be monitored by a direct arterial catheter 22 gauge inserted by the surgeon into the pulmonary artery, immediately after sternotomy, after aortic clamp removal, and 10 minutes after initiation of protamine infusion
Change in direct pulmonary artery systolic pressure (PASP) measured in mmHg | 10 minutes after initiation of protamine
  he pulmonary artery systolic pressure (PASP) will be monitored by a direct arterial catheter 22 gauge inserted by the surgeon into the pulmonary artery, immediately after sternotomy, after aortic clamp removal, and 10 minutes after initiation of protamine infusion

SECONDARY OUTCOMES:
• Lung ultrasound score. | beginning of surgery
  The sum of lung comets will produce a score reflecting the extent of LW accumulation. The lung ultrasound score will be obtained by scanning 12-rib interspaces with the probe longitudinally applied perpendicular to the wall. Each hemi-thorax will be divided in six areas: The sum of B-lines found on each scanning site (0: absence; 1: B7 lines: multiple B-lines 7 mm apart; 2: B3 lines: multiple B 3 mm apart; 3: consolidation) yields a score
Change in Lung ultrasound score | End of suregery
  The sum of lung comets will produce a score reflecting the extent of LW accumulation. The lung ultrasound score will be obtained by scanning 12-rib interspaces with the probe longitudinally applied perpendicular to the wall. Each hemi-thorax will be divided in six areas: The sum of B-lines found on each scanning site (0: absence; 1: B7 lines: multiple B-lines 7 mm apart; 2: B3 lines: multiple B 3 mm apart; 3: consolidation) yields a score

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Hefnawy, profesor, Study Chair — Cairo unuversity
Locations (1):
- Cairo University Pediatric Hospitals, Giza, الجيزة, Egypt

IPD SHARING:
Plan to Share IPD: No